CLINICAL TRIAL: NCT00114166
Title: A Randomized Phase II Evaluation of Topotecan (NSC #609699) Administered Daily x 5 Every 3 Weeks vs Weekly Topotecan in the Treatment of Recurrent Platinum-Sensitive Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Topotecan in Treating Patients With Recurrent Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0146Q; GOG-0146Q; CDR0000434848
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2014-05

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topotecan 1.25 mg/m2 IV days 1-5 of a 21 day cycle (Active Comparator): Topotecan 1.25 mg/m2 IV days 1-5 of a 21 day cycle until disease progression or adverse effects prohibit further therapy
  Interventions: Drug: topotecan hydrochloride
- Topotecan 4.0 mg/m2 IV day 1, 8 and 15 of a 28 day cycle (Active Comparator): Topotecan 4.0 mg/m2 IV day 1, 8 and 15 of a 28 day cycle until disease progression or adverse effects prohibit further therapy
  Interventions: Drug: topotecan hydrochloride

INTERVENTIONS:
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving topotecan in different dosing schedules may kill more tumor cells.

PURPOSE: This phase II trial is studying how well topotecan works in treating patients with recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of topotecan, in terms of frequency and duration of tumor response, in patients with recurrent platinum-sensitive ovarian epithelial, fallopian tube, or primary peritoneal cancer.
* Determine the nature and degree of toxicity of this regimen in these patients.

Secondary

* Determine the duration of progression-free survival and overall survival in patients treated with these regimens.
* Determine the effects of prognostic variables (i.e., initial performance status, age, and mucinous or clear cell histology) in patients treated with these regimens.

OUTLINE: This is a multicenter study.

Patients receive topotecan IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: Approximately 38-110 patients (19-55 per treatment arm) will be accrued for this study within 15-30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal cancer

  * Recurrent disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * At least 1 target lesion not in a previously irradiated field
* Received 1, and only 1, prior platinum-based chemotherapy regimen for primary disease containing carboplatin, cisplatin, or other organoplatinum compound

  * Initial treatment may have included high-dose, consolidation, or extended therapy administered after surgical or non-surgical assessment
  * Patients who have not received prior paclitaxel may receive a second regimen that includes paclitaxel
* Platinum-sensitive disease

  * Treatment-free interval* without clinical evidence of progressive disease for > 6 months after prior response to a platinum-based regimen NOTE: *Non-platinum maintenance or consolidation therapy is not included in calculation of the treatment-free interval
* Not eligible for a higher priority GOG protocol (i.e., any active phase III GOG protocol for the same patient population)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN
* Creatinine clearance > 40 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No sensory or motor neuropathy > grade 1
* No active infection requiring antibiotics
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 weeks since prior biologic or immunologic agents for the malignancy
* No more than 1 prior non-cytotoxic (biologic or cytostatic) regimen (e.g., monoclonal antibodies, cytokines, or small molecule inhibitors of signal transduction) for recurrent disease
* No concurrent cytokines during the first course of study treatment
* No concurrent pegfilgrastim

Chemotherapy

* See Disease Characteristics
* See Biologic therapy
* Recovered from prior chemotherapy
* No other prior cytotoxic chemotherapy for recurrent disease, including retreatment with initial chemotherapy regimen
* No prior topotecan

Endocrine therapy

* At least 1 week since prior hormonal therapy for the malignancy
* Concurrent hormone replacement therapy allowed

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy
* No prior radiotherapy to > 25% of marrow-bearing areas

Surgery

* Recovered from prior surgery

Other

* At least 3 weeks since other prior therapy for the malignancy
* No prior anticancer therapy that would preclude study treatment

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2005-01; Primary Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Herzog, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (78):
- United States (78):
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Woman's Hospital, Baton Rouge, Louisiana
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Jersey Shore Cancer Center at Jersey Shore University Medical Center, Neptune City, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Midtown Tulsa, Tulsa, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Harrington Cancer Center, Amarillo, Texas
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin

REFERENCES:
- [Result] Herzog TJ, Sill MW, Walker JL, O'Malley D, Shahin M, DeGeest K, Weiner SA, Mutch D, DeBernardo RL, Lentz SS. A phase II study of two topotecan regimens evaluated in recurrent platinum-sensitive ovarian, fallopian tube or primary peritoneal cancer: a Gynecologic Oncology Group Study (GOG 146Q). Gynecol Oncol. 2011 Mar;120(3):454-8. doi: 10.1016/j.ygyno.2010.11.008. Epub 2010 Dec 17. PMID 21168198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Regimen 1 (Topotecan 1.25 mg/m2) recruitment ended early due to lack of interest by institutions.
Groups:
- Regimen I (Topotecan 1.25 mg/m2): Regimen I Topotecan 1.25 mg/m2 IV days 1-5 of a 21-day cycle until disease progression or adverse effects prohibit further therapy
- Regimen II (Topotecan 4.0 mg/m2 ): Regimen II Topotecan 4.0 mg/m2 IV day 1, 8 and 15 of a 28-day cycle until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | Regimen I (Topotecan 1.25 mg/m2) | Regimen II (Topotecan 4.0 mg/m2 )
Started | 15 | 66
Completed | 15 | 65
Not Completed | 0 | 1
Not completed — Wrong primary | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Groups:
- Regimen II (Topotecan 4.0 mg/m2): Regimen II Topotecan 4.0 mg/m2 IV day 1, 8 and 15 of a 28-day cycle until disease progression or adverse effects prohibit further therapy
- Total: Total of all reporting groups
Arm/Group | Regimen I (Topotecan 1.25 mg/m2) | Regimen II (Topotecan 4.0 mg/m2) | Total
Number analyzed (Participants) | 15 | 65 | 80
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 2 | 5 | 7
  50-59 years | 3 | 29 | 32
  60-69 years | 4 | 17 | 21
  70-79 years | 5 | 12 | 17
  > 79 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 65 | 80
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 65 | 80
Cell Type [Number; unit: participants]
  Adenocarcinoma, Unspecified | 0 | 5 | 5
  Clear Cell Carcinoma | 1 | 1 | 2
  Endometrioid Adenocarcinoma | 0 | 2 | 2
  Mixed Epithelial Carcinoma | 1 | 5 | 6
  Undifferentiated Carcinoma | 0 | 1 | 1
  Serous Adenocarcinoma | 13 | 50 | 63
  Other Carcinoma | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response
Description: Response is measured according to Response Evaluation Criteria in Solid Tumors Criteria (RECIST v 1.0):
  Complete Response (CR) is disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart.
  Partial Response (PR) is at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD.
  Disease Progression is at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD or the appearance of new lesions within 8 weeks of study entry.
  Stable Disease is any condition not meeting the above criteria.
  Indeterminate is defined as having no repeat tumor assessments following initiation of study therapy for reasons unrelated to symptoms or signs of disease.
Time Frame: Every other cycle for the first 6 months, then every 3 months x2, then every 6 months until disease progression or study withdrawal
Population: Eligible and evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen I (Topotecan 1.25 mg/m2) | Regimen II (Topotecan 4.0 mg/m2)
Number analyzed (Participants) | 15 | 65
Participants
  Partial Response | 4 | 8
  Stable Disease | 8 | 32
  Increase Disease | 2 | 21
  Indeterminate | 1 | 4

2. Primary Outcome: Number of Participants With Adverse Effects (Grade 3 or Higher) as Assessed by Common Toxicity Criteria for Adverse Events Version 2.0
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Groups:
- Regimen I: Topotecan 1.25 mg/m2 IV days 1-5 of a 21-day cycle until disease progression or adverse effects prohibit further therapy
- Regimen II: Topotecan 4.0 mg/m2 IV day 1, 8 and 15 of a 28-day cycle until disease progression or adverse effects prohibit further therapy
Arm/Group | Regimen I | Regimen II
Number analyzed (Participants) | 15 | 65
Participants
  Leukopenia | 10 | 6
  Thrombocytopenia | 7 | 6
  Neutropenia | 14 | 18
  Anemia | 5 | 9
  Nausea/vomiting | 1 | 1
  Other Gastrointestinal | 1 | 0
  Neurologic | 0 | 1
  Constitutional | 1 | 2
  Cardiovascular | 1 | 0
  Infection | 1 | 2
  Musculoskeletal | 0 | 1
  Pulmonary | 1 | 2
  Pain | 0 | 4

3. Secondary Outcome: Reason Off Study Therapy
Time Frame: study entry through end of study treatment, up to 5 years
Population: Eligible and evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen I (Topotecan 1.25 mg/m2) | Regimen II (Topotecan 4.0 mg/m2)
Number analyzed (Participants) | 15 | 65
Participants
  Disease Progression | 9 | 47
  Refused further treatment | 3 | 7
  Toxicity as permitted | 3 | 2
  Other | 0 | 9

ADVERSE EVENTS:
Time Frame: All patients followed until disease progression or study withdrawal. In addition, following disease progression, patients will be monitored for delayed toxicity for a period of 5 years.
Arm/Group | Regimen I | Regimen II
Serious Adverse Events (participants affected / at risk) | 8/15 | 10/65
Other Adverse Events (participants affected / at risk) | 10/15 | 60/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen I (N=15) | Regimen II (N=65)
Neutrophils (Blood and lymphatic system disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1
Obstruction, Gi - Cecum (Gastrointestinal disorders) | 1 | 0
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Dehydration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 1 | 0
Inf W/Gr 3 Or 4 Anc: Bronchus (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Mood Alteration - Depression (Nervous system disorders) | 0 | 1
Pain: Back (General disorders) | 1 | 0
Pain: Abdominal Pain Nos (General disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen I (N=15) | Regimen II (N=65)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 0 | 3
Rhinitis (Immune system disorders) | 0 | 3
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Neutrophils (Blood and lymphatic system disorders) | 9 | 44
Platelets (Blood and lymphatic system disorders) | 8 | 38
Leukocytes (Blood and lymphatic system disorders) | 8 | 47
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 8 | 58
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 2
Ventricular Arrhythmia - Tachycardia (Cardiac disorders) | 0 | 1
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 0 | 3
S/N Arrhythmia: Atrial Tachycardia (Cardiac disorders) | 0 | 1
Hypertension (Cardiac disorders) | 0 | 7
Hypotension (Cardiac disorders) | 0 | 3
Inr (Vascular disorders) | 0 | 1
Ptt (Vascular disorders) | 0 | 2
Sweating (General disorders) | 1 | 5
Weight Gain (General disorders) | 0 | 3
Fever (General disorders) | 1 | 9
Weight Loss (General disorders) | 0 | 3
Rigors/Chills (General disorders) | 0 | 5
Fatigue (General disorders) | 8 | 46
Insomnia (General disorders) | 2 | 14
Nail Changes (Skin and subcutaneous tissue disorders) | 0 | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 5 | 19
Bruising (Skin and subcutaneous tissue disorders) | 0 | 5
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Skin and subcutaneous tissue disorders) | 1 | 1
Hand-Foot (Skin and subcutaneous tissue disorders) | 0 | 1
Hot Flashes (Endocrine disorders) | 0 | 3
Diabetes (Endocrine disorders) | 0 | 3
Flatulence (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Heartburn (Gastrointestinal disorders) | 2 | 8
Ulcer,gi - Stomach (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0
Distention (Gastrointestinal disorders) | 2 | 4
Taste Alteration (Gastrointestinal disorders) | 0 | 7
Incontinence, Anal (Gastrointestinal disorders) | 0 | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 0 | 5
Vomiting (Gastrointestinal disorders) | 4 | 12
Anorexia (Gastrointestinal disorders) | 2 | 16
Dehydration (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 5 | 29
Nausea (Gastrointestinal disorders) | 7 | 39
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 10
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 0 | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 0 | 2
Hemorrhage, Gi - Anus (Vascular disorders) | 0 | 1
Hemorrhage, Gi - Oral Cavity (Vascular disorders) | 0 | 1
Petechiae (Vascular disorders) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 0 | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 0 | 1
Inf Unknown Anc: Sinus (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Dental-Tooth (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 0 | 4
Infection - Other (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 0 | 2
Inf Unknown Anc: Bronchus (Infections and infestations) | 0 | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 0 | 3
Inf Unknown Anc: Catheter-Related (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 0 | 1
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 0 | 1
Edema: Limb (Blood and lymphatic system disorders) | 2 | 11
Edema: Head And Neck (Blood and lymphatic system disorders) | 1 | 0
Ast (Metabolism and nutrition disorders) | 0 | 9
Gfr (Metabolism and nutrition disorders) | 0 | 2
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 0 | 2
Cholesterol,serum High (Metabolism and nutrition disorders) | 0 | 1
Proteinuria (Metabolism and nutrition disorders) | 0 | 1
Creatinine (Metabolism and nutrition disorders) | 1 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 3
Alt (Metabolism and nutrition disorders) | 1 | 8
Alkaline Phosphatase (Metabolism and nutrition disorders) | 2 | 8
Bilirubin (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatremia (Metabolism and nutrition disorders) | 2 | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 2
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 0 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 20
Hypokalemia (Metabolism and nutrition disorders) | 1 | 11
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 10
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint-Function (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 6
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 0 | 5
Muscle Weakness - Extremity-Upper (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 1
Involuntary Movement (Nervous system disorders) | 0 | 1
Mood Alteration - Depression (Nervous system disorders) | 2 | 8
Mood Alteration - Anxiety (Nervous system disorders) | 0 | 7
Mood Alteration - Agitation (Nervous system disorders) | 0 | 1
Speech Impairment (Nervous system disorders) | 0 | 1
Cognitive Disturbance (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Confusion (Nervous system disorders) | 0 | 2
Memory Impairment (Nervous system disorders) | 0 | 4
Dizziness (Nervous system disorders) | 2 | 8
Neuropathy-Sensory (Nervous system disorders) | 3 | 26
Neuropathy-Motor (Nervous system disorders) | 0 | 3
Ocular/Visual - Other (Eye disorders) | 0 | 2
Watery Eye (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Blurred Vision (Eye disorders) | 2 | 4
Pain - Other (General disorders) | 1 | 4
Pain: Urethra (General disorders) | 0 | 1
Pain: Pelvis (General disorders) | 0 | 3
Pain: Chest /Thorax Nos (General disorders) | 1 | 5
Pain: Chest Wall (General disorders) | 1 | 1
Pain: Throat/Pharynx/Larynx (General disorders) | 0 | 2
Pain: Head/Headache (General disorders) | 1 | 11
Pain: Neck (General disorders) | 0 | 1
Pain: Extremity-Limb (General disorders) | 0 | 10
Pain: Back (General disorders) | 2 | 9
Pain: Joint (General disorders) | 0 | 5
Pain: Bone (General disorders) | 0 | 2
Pain: Lymph Node (General disorders) | 0 | 1
Pain: Kidney (General disorders) | 1 | 0
Pain: Pain Nos (General disorders) | 0 | 1
Pain: Oral Cavity (General disorders) | 0 | 1
Pain: Dental/Teeth/Peridontal (General disorders) | 0 | 2
Pain: Abdominal Pain Nos (General disorders) | 3 | 16
Pain: Tumor (General disorders) | 0 | 1
Pain: Muscle (General disorders) | 1 | 2
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 13
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 21
Cystitis (Renal and urinary disorders) | 0 | 3
Urinary Retention (Renal and urinary disorders) | 0 | 2
Obstruction, Gu - Ureter (Renal and urinary disorders) | 0 | 1
Incontinence, Urinary (Renal and urinary disorders) | 0 | 2
Bladder Spasm (Renal and urinary disorders) | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 2 | 1
Libido (Reproductive system and breast disorders) | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No